CLINICAL TRIAL: NCT00188279
Title: Minimum Dose Computed Tomography of the Thorax for Follow-up in Patients With Resected Lung Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-0051-C
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: ct; scan; lung; follow-up
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MnDCT (Experimental)
  Interventions: Procedure: Minimum Dose Computed Tomography (MnDCT) scan

INTERVENTIONS:
Procedure: Minimum Dose Computed Tomography (MnDCT) scan — Minimum Dose Computed Tomography (MnDCT) scan at regular follow up intervals for up to 5 years post-operatively.

SUMMARY:
This study is designed to help decide whether a CAT scan performed at a very low dose of radiation (Minimum dose CT scan) is better than a Chest X-Ray in detecting recurrence of lung cancer in the chest (after surgery).

DETAILED DESCRIPTION:
Lung Carcinoma is expected to kill 18,900 men and women in Canada in 2004. This is more than the combined total for the next three common cancers. The most important factor that determines patient survival is the stage of disease at presentation. Surgical resection is the best chance of cure. However, patients who undergo lung resection with curative intent have a significant incidence of a second lung cancer at 2% per year and a recurrence rate of 38% at 5 years. The current follow-up of these patients relies on periodic physical examination and chest radiography(CXR). However, CXR is insensitive in the detection of lung nodules when compared to standard Computed Tomography of the thorax (SDCT). Computed Tomography detects smaller lung nodules than CXR however, the radiation dose from a SDCT is roughly equivalent to 20 CXR examinations. Screening studies using Low Dose CT of the Thorax (LDCT) in subjects at high risk for lung cancer have demonstrated that LDCT detects three times as many nodules as CXR and four times as many primary lung cancers at one-third the dose of SDCT. Phantom and clinical work with LDCT performed at UHN/MSH suggests that a further reduction in radiation dose (Minimum Dose CT -MnDCT) is possible for nodule detection. Minimum dose CT is performed at a dose one sixth of a SDCT.In addition, if MnDCT is confirmed to be a more sensitive nodule detection technique, it could be used to

1. Increase the interval between repeat out-patient assessment and thereby 2. Reduce the overall cost of surveillance and inconvenience to the patient and 3. Free up clinic time for the surgeon to review more patients and reduce waiting lists

ELIGIBILITY:
Inclusion Criteria:

* lung cancer patients undergoing resection with intent to cure

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2005-06-21; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Detection of local recurrent disease | 5 years
Evaluate the incidence and significance of sub-5mm lung nodules in this patient population | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada